CLINICAL TRIAL: NCT01153594
Title: Early Re-Intervention (ERI) Experiment 2
Brief Title: Early Re-Intervention Experiment 2
Acronym: ERI2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Michael L. Dennis, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERI-2; 5R37DA011323 (NIH)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Substance Use Disorders
Keywords: Substance Use Disorders; Relapse; Recovery; Disease Management; Long term outcomes; Addiction Treatment
MeSH Terms: conditions — Substance-Related Disorders; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recovery Management Checkups (RMC) (Experimental): Participants in the RMC group are interviewed quarterly. When they were found to be in need of treatment, the participant was transferred from the interviewer to a linkage manager to receive the intervention (described next). They were also able to re-enter treatment on their own and naturally cycle through multiple periods of substance use, treatment, incarceration and recovery.
  Interventions: Behavioral: Recovery Management Checkups (RMC)
- Control Group (No Intervention): Participants in the control group are interviewed quarterly. While they do not receive any active intervention from the research team, they are able to re-enter treatment on their own and naturally cycle through multiple periods of substance use, treatment, incarceration and recovery.

INTERVENTIONS:
Behavioral: Recovery Management Checkups (RMC) — After interviewers completed the quarterly research interview and determined participants' eligibility and need for early re-intervention, they transferred RMC participants who were eligible and in need to a Linkage Manager. Using motivational interviewing, the Linkage Manager: a) provided feedback to participants regarding their current substance use and related problems, b) discussed implications of managing addiction as a chronic condition, c) discussed treatment barriers and solutions, d) assessed and discussed level of motivation for treatment, e) scheduled treatment appointments, f) accompanied participants to treatment intake and stayed through the process, and g) implemented Engagement and Retention Protocol during the 14 days of treatment
  Arms: Recovery Management Checkups (RMC)

SUMMARY:
The objective of this study was to evaluate the relative effectiveness of quarterly Recovery Management Checkups (RMC) on long-term outcomes of adult chronic substance users over 4 years.

DETAILED DESCRIPTION:
CONTEXT: While drug abuse is the 10th leading cause of mortality in the US, the disorder remains an orphan of the public health care system. Unlike cancer, diabetes, and other chronic diseases, the detection, re-emergence, and progression of which we have learned to respond with aggressively timed monitoring and interventions, drug abuse remains isolated from adoption into the "chronic condition" model of care.

OBJECTIVES AND HYPOTHESES: The objective of this study was to evaluate the relative effectiveness of quarterly checkups on long-term outcomes of adult chronic substance users over 4 years. Relative to participants randomly assigned to the control group, we predicted that RMC participants would: H1) return to treatment sooner, H2) receive more treatment, H3) decrease substance use, and H4) increase days of abstinence.

METHOD: Participants were recruited from sequential intakes at the largest addiction treatment agency in Illinois between February and April of 2004. Inclusion criteria were: any substance use in the past 90 days and any past-year symptoms of substance use disorders. For logistical reasons, participants were excluded if they were: under 18, lived or planned to move outside Chicago within 12 months, sentenced to a confined environment most of the next 12 months, mandated to treatment because of a driving under the influence offense, were not fluent in English or Spanish, or were cognitively unable to provide informed consent. To evaluate efficacy of quarterly Recovery Management Checkups (RMC) on treatment reentry and substance use, 446 adults (88% with dependence criteria) were randomly assigned quarterly RMCs, or, an outcome monitoring only control group and followed quarterly for 4 years (94% completion).

INTERVENTION. After interviewers completed the quarterly research interview and determined participants' eligibility and need for early re-intervention, they transferred RMC participants who were eligible and in need to a Linkage Manager. Using motivational interviewing, the Linkage Manager: a) provided feedback to participants regarding their current substance use and related problems, b) discussed implications of managing addiction as a chronic condition, c) discussed treatment barriers and solutions, d) assessed and discussed level of motivation for treatment, e) scheduled treatment appointments, f) accompanied participants to treatment intake and stayed through the process, and g) implemented Engagement and Retention Protocol during the 14 days of treatment. Detailed procedures and forms are available in the RMC manual(Scott & Dennis, 2003; http://www.chestnut.org/LI/downloads/Scott_&_Dennis_2003_RMC_Manual-2_25_03.pdf ).

OUTCOME MEASURES: Days to first treatment, days of treatment, successive quarters of needing treatment, number of substance problem months, days of abstinence.

ELIGIBILITY:
Inclusion Criteria:

* any substance use in the past 90 days
* any past-year symptoms of substance use disorders.

Exclusion Criteria:

* under 18
* lived or planned to move outside Chicago within 12 months
* sentenced to a confined environment most of the next 12 months
* mandated to treatment because of a driving under the influence offense
* were not fluent in English or Spanish
* were cognitively unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2004-02; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Time to First Alcohol or Drug Treatment Re-Entry | Quarterly from random assignment until month 48
  Days to readmission was calculated as the number of days from the date of the quarterly follow-up interview where the client first reported being in need of treatment (see below) to the date of the first subsequent intake to alcohol or other drug treatment following that interview.

SECONDARY OUTCOMES:
Any Treatment Re-Entry | Quarterly from random assignment until month 48
  Whether the person re-entered treatment between the point of randomization (at 3 months) and last observation.
Times Re-entered Treatment Time Frame | Quarterly from random assignment until month 48 Description:
  Number of times client re-entered treatment between randomization and the last observation.
Total Days of Treatment | Quarterly from random assignment until month 48
  Based on the sum of days an individual received outpatient, intensive outpatient, residential, or inpatient treatment reported at each interview for a given period.
Quarters with 7 days Outpatient or 14 days Residential | Quarterly from random assignment until month 48
  The number of quarters a participant received treatment at least 7 days of outpatient or 14 days of residential treatment, regardless of whether it is due to retention, step down or readmission.
Quarters Needing Treatment | Quarterly from random assignment until month 48
  Defined as a participant living in the community (vs. in incarcerated) who was not already in treatment and had been intoxicated or used alcohol or drugs on 13 or more of the past 90 days; had any symptoms of abuse, dependence, or withdrawal in the past month; or currently felt the need to return to treatment. Within quarter these criteria for need are internally consistent (alpha=.85) and the average person in need endorsed 3.3 of 6 of the items (80% endorsed 2 or more).
Successive Quarters Needing Treatment | Quarterly from random assignment until month 48
  The number of quarters in which the individual started and ended the period "in need of treatment" (see definition above) where missing data were replaced with status at prior wave.
Substance Problem x Months | Quarterly from random assignment until month 48
  Count of 16 past-month item related to weekly use, hiding using, complaints about use, 4 symptoms of abuse, 7 symptoms of dependence, substance induced health or mental health asked for the month before each quarterly interview times 3 and summed over observations; using mean score for any missing observations.
Total Days of Abstinence | Quarterly from random assignment until month 48
  Sum of days abstinent from alcohol or other drugs in months 4 to 48 (max=1350 days); using the mean days per quarter for any missing observations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Dennis, Ph.D., Principal Investigator — Chestnut Health Systems; Christy K Scott, Ph.D., Principal Investigator — Chestnut Health Systems
Locations (1):
- Chestnut Health Systems, Chicago, Illinois, United States

REFERENCES:
- [Background] Scott CK, Sonis J, Creamer M, Dennis ML. Maximizing follow-up in longitudinal studies of traumatized populations. J Trauma Stress. 2006 Dec;19(6):757-69. doi: 10.1002/jts.20186. PMID 17195975
- [Background] Dennis M, Scott CK. Managing addiction as a chronic condition. Addict Sci Clin Pract. 2007 Dec;4(1):45-55. doi: 10.1151/ascp074145. PMID 18292710
- [Result] Rush BR, Dennis ML, Scott CK, Castel S, Funk RR. The interaction of co-occurring mental disorders and recovery management checkups on substance abuse treatment participation and recovery. Eval Rev. 2008 Feb;32(1):7-38. doi: 10.1177/0193841X07307532. PMID 18198169
- [Result] Scott CK, Dennis ML. Results from two randomized clinical trials evaluating the impact of quarterly recovery management checkups with adult chronic substance users. Addiction. 2009 Jun;104(6):959-71. doi: 10.1111/j.1360-0443.2009.02525.x. Epub 2009 Mar 13. PMID 19344441
- [Derived] McCollister KE, French MT, Freitas DM, Dennis ML, Scott CK, Funk RR. Cost-effectiveness analysis of Recovery Management Checkups (RMC) for adults with chronic substance use disorders: evidence from a 4-year randomized trial. Addiction. 2013 Dec;108(12):2166-74. doi: 10.1111/add.12335. Epub 2013 Oct 9. PMID 23961833